CLINICAL TRIAL: NCT05258851
Title: Ceftazidime-Avibactam Versus Colistin in Critically Ill Patients With Carbapenem-Resistant Enterobacteriaceae Infections (AVI-ICU): A Non-Inferiority Randomized Clinical Trial
Brief Title: Ceftazidime-Avibactam Use in Critically Ill Patients With Carbapenem-Resistant Enterobacteriaceae Infections
Acronym: AVI-ICU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties encountered in the recruitment process and slow enrollment. The study was not terminated due to any safety issues or concerns.
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Zainab Alduhailib, Critical Care Medicine Consultant, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAC#2211247
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection
Keywords: Carbapenem-Resistant Enterobacteriaceae; Critically ill; Ceftazidime-avibactam; Colistin
MeSH Terms: conditions — Critical Illness | interventions — avibactam, ceftazidime drug combination; Colistin

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, parallel-group, stratified, non-inferiority randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ceftazidime-avibactam (Experimental): Ceftazidime-avibactam 2.5 grams intravenous (IV) every 8 hours infused over two hours for a duration of 7-14 days, with dose adjustment for renal impairment according to the FDA prescribing information. Patients who have a positive Xpert Carb-R screening test or culture for CRE with metallo-beta-lactamases will receive aztreonam added to ceftazidime-avibactam.
  Interventions: Drug: Ceftazidime-avibactam
- Colistin (Active Comparator): Colistin (9-million-unit loading dose IV followed with 9 million units IV daily divided into 3 doses), for 7 to 14 days. Patients with renal impairment will receive antibiotics with adjusted doses based on their glomerular filtration rate or the use and type of renal replacement therapy according to the 2019 International Consensus Guidelines for the Optimal Use of the Polymyxins.
  Interventions: Drug: Colistin

INTERVENTIONS:
Drug: Ceftazidime-avibactam — Experimental
  Arms: Ceftazidime-avibactam
Drug: Colistin — Control
  Arms: Colistin

SUMMARY:
Carbapenem-Resistant Enterobacteriaceae (CRE) infections are a growing national and international challenge in healthcare settings. This is not only due to the rapid spread of resistance and paucity of options of targeted-antimicrobial agents, but also owing to the high mortality of patients infected with CRE reaching up to 50% as per the Centers of Disease Control and Prevention.

Colistin-based combination regimens have been the mainstay for treating CRE-related infections. Ceftazidime-avibactam is a beta-lactamase inhibitor combination, a novel antibiotic, which recently showed a better clinical and microbiological cure against CRE along with the potential to reduce mortality and nephrotoxicity in comparison to colistin-based regimens in observational studies. However, randomized clinical trials are lacking.

This non-inferiority randomized controlled study aims to assess the efficacy and safety of ceftazidime-avibactam-based regimens in critically ill patients with CRE infections in comparison to colistin-based regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years.
2. Admitted to an intensive care unit (ICU).
3. Patients with hospital-acquired pneumonia (HAP) or ventilator-associated pneumonia (VAP), complicated urinary tract infection (cUTI), bacteremia, complicated intraabdominal infection (cIAI), and complicated skin and soft tissue infection (cSSTI).
4. Confirmed infection with CRE, based on a culture and sensitivity obtained within the past 72 hours of study enrollment.
5. Suspected CRE infection according to one of the following: (1) positive Xpert Carba-R test screening for blaKPC or blaOXA-48 or blaNDM or blaVIM or blaIMI assessed on the admission to the ICU, (2) positive culture for CRE obtained within 3 months from time of enrollment.

Exclusion Criteria:

1. Acute Physiology and Chronic Health Evaluation II (APACHE II) score more than 30
2. known significant hypersensitivity reaction to beta-lactam antibiotics or colistin
3. Positive culture for Stenotrophomonas maltophilia or Acinetobacter baumannii within the current hospitalization.
4. Patients received the study intervention or control for more than 24 hours before the intended randomization.
5. Patient/substitute decision-maker or caring physician's refusal to enroll in the study.
6. Patient with concomitant suspected or confirmed meningitis.
7. Pregnancy.
8. Cystic fibrosis.
9. Patients with Do Not Attempt to Resuscitate (DNAR) code status.
10. Prior knowledge that the index CRE pathogen was resistant to colistin (MIC >2 μg/ml) or ceftazidime-avibactam (MIC > 8 μg/ml) before randomization.
11. Objective clinical evidence for any of the following infections that necessitate study therapy for >14 days: endovascular infection, including endocarditis, osteomyelitis, prosthetic joint infection, meningitis, and/or other central nervous system infections

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days from randomization
  Death

SECONDARY OUTCOMES:
14-day mortality | 14 days from randomization
  Death
Number of patients with clinical success at end of therapy (EOT) at day 7-14 from randomization and test of cure (TOC) 7 days after completion of treatment | EOT at 7-14 days from randomization and TOC 7 days after completion of treatment
  Defined as:
  1- Alive, fever or hypothermia resolution, WBC counts normalization, hemodynamic stability with MAP ≥65 mmHg without vasopressors support.
  1. For HAP or VAP: 1+ improving respiratory status including improving PaO2/FiO2 ratio from baseline, decreasing FiO2 and PEEP or extubation or source control for empyema.
  2. For bloodstream infection: 1+ documented two negative blood cultures with source removal if applicable.
  3. For complicated intra-abdominal infection: 1+ resolution or decreasing size of intra-abdominal collections with source control if applicable.
  4. For complicated skin and soft tissue infection: 1+ resolution of signs and symptoms plus surgical drainage or debridement if applicable.
  5. For complicated urinary tract infection: 1+ resolution of signs and symptoms and source removal if applicable.
Number of patients with microbiological response at the EOT at days 7-14 from randomization and TOC 7 days after completion of treatment | EOT at 7-14 days from randomization and TOC 7 days after completion of treatment
  Defined as:
  1. Eradication (successful microbiological response): Baseline pathogen no longer present in the culture(s) that indicated the use of study drugs.
  2. Presumed eradication (successful microbiological response): Patient deemed a clinical cure as assessed by the adjudication committee at EOT and TOC, and repeat culture that indicated enrollment in the study is not available.
  3. Persistence (failure of microbiological response): Presence of baseline pathogen in the culture that indicated the use of study drugs.
  4. Presumed persistence (failure of microbiological response): Patients deemed a clinical failure as assessed by the adjudication committee at EOT and TOC, and specimen is not available.
  5. Indeterminate: Any culture that cannot be classified into one of the above categories, or the patient was an indeterminate clinical response and no cultures were taken.
Time to weaning from mechanical ventilation at day 28 | 28 days from randomization
  Number of days not receiving mechanical ventilation
Requirement for renal replacement therapy at day 28 | 28 days from randomization
  New start of renal replacement therapy
Intensive care unit (ICU) length of stay, censored at 28 days | 28 days from randomization
  Duration of stay inside the ICU
Days alive and out of the ICU, censored at 28 days | 28 days from randomization
  Number of days alive and outside the ICU
Drug-related adverse events | 28 days from randomization
  Acute kidney injury, seizures, leukopenia, thrombocytopenia, allergic reaction, diarrhea, clostridium difficile infection.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Al Duhailib, Principal Investigator — King Faisal Specialist Hospital & Research Center; Hakeam Hakeam, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No